CLINICAL TRIAL: NCT05096195
Title: Denosumab for the Prevention of Fragility Fractures in Hemodialysis: a Pilot Study for an Innovative, Randomized-controlled Trial, Embedded in Routine Care
Brief Title: PRevEnting FracturEs in REnal Disease - 1
Acronym: PREFERRED-1
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: ICES (Industry); Academic Medical Organization of Southwestern Ontario (Other); Western University (Other); The Kidney Foundation of Canada (Other)
Responsible Party: Principal Investigator, Kristin Clemens, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3638
Record Dates: First submitted 2021-09-21; First posted 2021-10-27 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Kidney Diseases; Dialysis; Complications; Fragility Fracture; Chronic Kidney Disease-Mineral and Bone Disorder
Keywords: Pilot Study; Fracture; denosumab; hemodialysis
MeSH Terms: conditions — Kidney Diseases; Chronic Kidney Disease-Mineral and Bone Disorder; Fractures, Bone | interventions — Denosumab; Calcium

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): 60 mg of denosumab (Prolia) will be administered every 6 months over a 15 - month period. Monitoring of serum calcium and phosphate will occur and bloodwork will be drawn for 7 weeks following each denosumab injection. Correction of vitamin D deficiency (if required), the adjustment of calcium dialysate and the provision of intravenous (IV) or oral (po) calcitriol/calcidiol will be administered as needed following each denosumab injection as described in the Beside Protocol. Once the study monitoring period is over, serum calcium monitoring and management will occur as per routine care in the dialysis centre. All intervention activities will occur during regularly scheduled hemodyalisis sessions.
  Interventions: Drug: Denosumab 60 mg/ml; Other: Calcium and vitamin D prophylaxis; Diagnostic Test: Monitoring of post-injection calcium and phosphate
- Usual care (No Intervention): Usual care participants will continue to receive the typical standard of care in their dialysis unit which includes their routine dialysis monitoring and bloodwork. They will not receive denosumab, calcium and vitamin prophylaxis. There will be no extra monitoring or bloodwork.

INTERVENTIONS:
Drug: Denosumab 60 mg/ml — Details described in intervention arm/group description section.
  Other Names: Prolia
  Arms: Intervention
Other: Calcium and vitamin D prophylaxis — Details described in intervention arm/group description section.
  Arms: Intervention
Diagnostic Test: Monitoring of post-injection calcium and phosphate — Details described in intervention arm/group description section.
  Arms: Intervention

SUMMARY:
PREFERRED-1 is a pilot study designed to determine the feasibility of a large randomized, pragmatic, open-label, comparative-effectiveness trial of denosumab for the prevention of fragility fractures in people receiving hemodialysis. The pilot study will enroll at least 60 patients from across at least 6 different hemodialysis centres in Ontario, Canada. Patients on outpatient maintenance hemodialysis at high risk of fragility fracture, will be randomized 1:1 to a denosumab care pathway vs. usual care.

Primary outcomes include recruitment feasibility and treatment adherence. Secondary outcomes include safety and participant satisfaction with our protocol and processes.

DETAILED DESCRIPTION:
Despite a fragility fracture risk that is >5-fold higher than those without chronic kidney disease (CKD), there is a lack of evidence on how to prevent fracture in patients on hemodialysis. Medications known to prevent fragility fracture in other populations, are either contraindicated in dialysis, or associated with severe side effects.

Denosumab (Prolia) is one of the only Health Canada approved medications for fragility fracture prevention across the CKD stages. While small clinical trials inclusive of hemodialysis patients have noted that denosumab improves bone mineral density and reduces bone turnover, whether this treatment effectively and safely prevents fragility fracture in this population still remains unclear.

Instead of conducting an expensive traditional RCT where results might fail to apply to the "real-world", the study will embed a trial of denosumab into routine care. The intervention will be delivered by healthcare staff. Participants will be closely followed at the dialysis unit where the participant has dialysis treatments. Baseline characteristics and outcomes will be captured using routine care data including administrative health data.

The overarching aim of the PREFERRED Program is to determine whether a denosumab care pathway vs. usual care (i.e., non-use of denosumab) alters the risk of fragility fracture in patients receiving in-centre hemodialysis. PREFERRED-1 is a pilot study that will inform the feasibility of conducting a large-scale, efficiently run, randomized-controlled trial in Canada to test whether denosumab reduces the risk of fragility fracture in patients receiving hemodialysis. The goal is to understand if individual level recruitment is feasible and timely, and if the intervention is acceptable to patients.

The objectives of PREFERRED-1 are to:

1. Examine whether streamlined methods of enrollment can facilitate recruitment across multiple centres in a timely way;
2. Demonstrate good adherence with the trial protocol and examine whether well-received by participants;
3. Ensure that participants are adherent with treatment assignment (i.e., intervention group to denosumab, minimal cross-over to denosumab in usual group);
4. Confirm there are no 'signals' of unmanageable harm (i.e. hypocalcemia) that would prevent testing of our intervention on a larger scale.

PREFERRED-1 will be deemed a success if:

* The study can randomly allocate at least 60 patients from at least 6 hemodialysis centres within 6-months of the trial being activated at each centre.
* Demonstrate that patients randomly allocated to denosumab receive over 90% of the scheduled injections at 0, 6 and 12 months
* Patients randomly allocated to no denosumab (i.e. usual care) do not receive a prescription for denosumab.

This "high-risk" innovative pragmatically approached trial focused on better treatments for fracture prevention in those with kidney disease will

1. inform transformational change in the care of real-world patients;
2. produce essential knowledge to safely prevent fracture in patients with kidney disease, and the associated costs to the healthcare system;
3. foster the conduct of collaborative, multidisciplinary care for those with complex kidney disease.

ELIGIBILITY:
Inclusion criteria:

* Treating nephrologist/nurse practitioner in the dialysis unit deems that a prescription for study drug (denosumab) will be safe/reasonable in the potential participant.
* Age ≥40 years
* Access to denosumab through provincial drug benefits (i.e. evidence of receiving outpatient prescription medications through the Ontario Drug Benefits Program, Ontario Disability Support Program)
* Baseline albumin-corrected serum calcium ≥2.15 mmol/L, PTH ≥15 pmol/L (or 2-9x the upper limit of normal for the local laboratory).
* High risk of fragility fracture defined by: a) ≥15% 10-year risk of major osteoporotic fracture or >3% 10-year risk of hip fracture (using the World Health Organization's Fracture Risk Assessment Tool which is validated in hemodialysis),OR b) a prior history of hip or vertebral fracture (where the later could have been asymptomatic and only observed radiographically), OR c) two or more fragility fractures of the humerus, wrist, and/or pelvis (e.g. 2 humerus fractures, humerus and wrist fracture).43

Exclusion criteria:

* Expected to recover kidney function, stop hemodialysis, pursue palliative care, or transfer to home or peritoneal dialysis within 12 months (as assessed by a health professional).
* Expected to start IV bisphosphonates (i.e. pamidronate or zoledronic acid).
* Current use of cinacalcet (Sensipar).
* Current use of an osteoporosis medication including:

  * Denosumab
  * Bisphosphonates
  * Alendronate (Fosavance or Fosamax)
  * Risedronate (Actonel or Actonel DR)
  * Zoledronic acid (Aclasta) or Pamidronate
  * Raloxifene (Evista)
  * Oral or conjugated estrogen
  * Topical, oral or injectable testosterone (Androgel, Testim, Fortesta, Androderm, testosterone enanthate and testosterone cypionate)
  * Teriperatide (Forteo)
  * Romosozumab (Evenity)
  * Calcitonin (Calcimar)
* Of childbearing status
* History of femur fracture attributed to osteoporosis medication use (i.e. midshaft femoral fracture or atypical femoral fracture)
* Major dental surgery planned within the next 6 months (e.g. root canal).
* Known allergy or intolerance to denosumab.
* Expected to receive a parathyroidectomy for hyperparathyroidism in the next 12 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 26 weeks
  Number or N (%) of participants randomly allocated within 26 weeks of trial initiation at each centre.
Adherence to study intervention | 15 months
  Number (%) of participants randomized to the intervention who received >90% of their scheduled treatments to study end.
Adherence to usual care | 15 months
  Number (%) of participants randomized to usual care who received no prescription for denosumab to study end.

SECONDARY OUTCOMES:
Treatment-related hypocalcemia as assessed by CTCAE v4.0 | within 7 weeks following denosumab injection
  N (%) with hypocalcemia and symptomatic hypocalcemia [graded according to common terminology criteria for adverse events v 4.0 criteria (Grade 2, albumin-corrected serum calcium 1.75 to 1.99 mmol/L, Grade 3, 1.5 to 1.74 mmol/L, Grade 4, serum calcium <1.5 mmol/L)] within 7 weeks of denosumab. Symptomatic hypocalcemia will be defined by a calcium <2.00 mmol/L in the presence of new muscle cramps or paresthesia.
Mean change in serum calcium | 7 weeks following denosumab injection
  Mean change in serum calcium from baseline to 7 weeks post injection
Median change in serum calcium | 7 weeks following denosumab injection
  Median change in serum calcium from baseline to 7 weeks post injection
Mean change in parathyroid hormone | 7 weeks following denosumab injection
  Mean change in parathyroid hormone from baseline to 7 weeks post injection
Median change in parathyroid hormone | 7 weeks following denosumab injection
  Median change in parathyroid hormone from baseline to 7 weeks post injection
Fragility fracture | 15 months
  N (%) with hospital encounter for fragility fracture of the hip, vertebrae, humerus, wrist, or pelvis at 15 months
Satisfaction with E-Platform and E-Consent Process | 15 months
  Patient satisfaction with e-platform, and e-consent process. (Likert Scale with 1=not satisfied to 5=very satisfied)
Satisfaction with intervention | 15 months
  Patient satisfaction with intervention (Likert Scale with 1=not satisfied, 5=very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin K Clemens, MD, MSc, Principal Investigator — St. Joseph's Health Care London
Locations (6):
- Canada (6):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Huron Perth Healthcare Alliance - Stratford General Hospital, Stratford, Ontario
  - St. Michaels Hospital, Toronto, Ontario
  - Woodstock Hospital, Woodstock, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clemens KK, Cowan A, Dixon S, Naylor K, Weir MA, Thain J, Khan T, Silver S, Molnar AO, Sultan N, Holden RM, Hiremath S, Wald R, Kitchlu A, Arnold J, Field B, Garg AX. PRevEnting FracturEs in REnal Disease-1 (PREFERRED-1): protocol for a pilot study of a pragmatic, randomised controlled trial of denosumab for the prevention of fragility fractures in haemodialysis. BMJ Open. 2025 Sep 10;15(9):e097195. doi: 10.1136/bmjopen-2024-097195. PMID 40935429